CLINICAL TRIAL: NCT06044545
Title: The Effect of Web Based Pregnancy Preparation Education Structured According to the Health Promotion Model in the Preconceptional Period on Women's Knowledge Attitude and Health Behaviors
Brief Title: Effect Web Based Pregnancy Preparation Education According to Health Promotion Model in Preconceptional Period on Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Ebru BOZCU, Instructor, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ebru1
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Health Promotion
Keywords: Preconceptional Period Health Promotion Pregnancy Education

STUDY DESIGN:
Intervention Model Description: A total of 84 people, 42 in the experimental group and 42 in the control group, will be included in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web Based Pregnancy Preparation Education Group (Experimental): Web Based Pregnancy Preparation Education Structured According to the Health Promotion Model Knowledge Attitude and Health Behaviors
  Interventions: Diagnostic Test: Web Based Pregnancy Preparation Education Structured According to the Health Promotion Model Knowledge Attitude and Health Behaviors
- Control Group (No Intervention): No action will be taken.

INTERVENTIONS:
Diagnostic Test: Web Based Pregnancy Preparation Education Structured According to the Health Promotion Model Knowledge Attitude and Health Behaviors — With this research, according to the "health promotion model" for the care that should be taken during the preconceptional period (pre-pregnancy) of women who are not yet pregnant, who will marry soon and who are considering pregnancy.
  It is thought that they will gain knowledge, increase their awareness and develop positive health behaviors with the "web-based pregnancy preparation training". In data collection; "Introductory Characteristics Form", "Preconceptional Knowledge and Attitudes Scale", "Preconception Health Behaviours Scale" will be used.
  Arms: Web Based Pregnancy Preparation Education Group

SUMMARY:
Preconceptional care is a very important preventive health service that gives couples the opportunity to prepare for a healthy pregnancy in a physically and psychologically healthy way, aims to identify and minimize the risks that may be present to the mother and fetus. Although preconceptional care is recommended for all couples of reproductive age, it is not at the desired level both in the world and in our country. In the literature, it is seen that the existing knowledge of individuals is insufficient, care is not provided for this period, and research revealing the knowledge and attitudes of individuals is very insufficient. It is thought that if the individuals in the society are informed about this issue and awareness is raised, the rate of benefiting from preconceptional care and counseling services will increase.

One of the important components of preconceptional counseling is health education. Health education aims to increase the knowledge of individuals, to create awareness and thus to gain positive health behavior. The Health Promotion Model enables individuals to make behavioral changes to create a healthy lifestyle. Based on this, this research has been planned in order to determine the effect of web-based pregnancy preparation education structured according to the health improvement model in the preconceptional period on women's knowledge, attitudes and health behaviors.

DETAILED DESCRIPTION:
One of the global health goals is to improve maternal health and reduce child mortality. In order to reduce maternal and newborn diseases and deaths, it is necessary to focus on preconceptional health. Preconceptional care aims to prepare individuals for pregnancy, to maintain and result in a healthy pregnancy, and to ensure that future generations are composed of healthier individuals. It is important to provide the necessary education, care and counseling to women in the preconception period in achieving these goals. The World Health Organization states that initiatives taken after pregnancy occur are quite late in reducing the risks to the mother and newborn. For this reason, it is necessary to take the necessary steps during the preconceptional period in order to create the highest level of impact on health outcomes.

When evaluated in general, nowadays; preconceptional care services and the rate of benefiting from these services are low all over the world, including many developed countries. For this reason, an important part of women today she still continues to conceive with preventable risks. It is stated in the literature that the proportion of those who have heard about the concept of preconceptional care and counseling is low; knowledge and positive behaviors related to preconceptional care are insufficient. In the literature, it has been determined that especially young, illiterate women or women living in poor areas do not have adequate access to pre-pregnancy, pregnancy and birth services. From this point of view, it is necessary to ensure the awareness of society about the preconceptional period and to conduct studies on the subject. It is thought that if the individuals in the society are informed about this issue and awareness is raised, the rate of benefiting from preconceptional care and counseling services will increase.

Education is an important component of preconceptional counseling. Health education is a combination of learning experiences designed to increase individuals' knowledge, create positive attitudes and improve their health. The main purpose of education is to first create awareness (positive attitude) by providing information and to develop correct behavior or change wrong behavior. The Health Promotion Model, on the other hand, provides individuals to make behavioral changes to create a healthy lifestyle. This research has been planned in order to determine the effect of web-based pregnancy preparation education structured according to the health improvement model in the preconceptional period on women's knowledge, attitudes and health behaviors.

Material and Method: This study is a randomized controlled trial. The research is planned to be conducted with women who applied for marriage to the Marriage Officer of Erzurum Metropolitan Municipality Social Services Department between February 2023 and February 2025. The sample number of the study was calculated using the G*Power 3.1.9.7 program. In the calculation, a sample calculation was performed for the t-test in independent groups (The Independent Samples T-Test) by taking into account the research design with 2 groups (Experimental Group, Control Group) and 2 measurements (pre-test - post-test). In the calculation made, the effect size was calculated as 0.80 (d = 0.80), 5% margin of error (α = 0.05) and 95% power (1-β = 0.95) and the number of samples for each group was calculated as 35. Considering the possibility of data loss, the number of samples in each group was increased by approximately 20% and determined as 42 people. In total, 84 women who applied for marriage were included in the sample.

In the collection of research data the introductory features form created by the researcher, "Preconceptional Knowledge and Attitudes Scale", "Preconception Health Behaviours Scale" will be used. In the evaluation of the data, SPSS package program will be used. Statistical significance level p<0.05 will be accepted as.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being literate in Turkish
* Never been pregnant
* Pregnancy in the last year plan
* Being able to use a computer
* Computer or mobile phone at home have a phone and internet connection

Exclusion Criteria:

* Questionnaire and/or scales incomplete answer
* Withdrawing from research
* Being pregnant

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Preparation for Pregnancy in the Preconceptional Period
Enrollment: 84 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2023-10-20 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Pre-Test Data Collection | Time frame: One or two months
  The pre-test data of the research will be collected by the researcher between September 2023 and October 2023, in line with the voluntariness of the women who applied to the Marriage Registry Office of the Erzurum Metropolitan Municipality Social Services Department for marriage. In collecting data, people in the experimental and control groups; "Introductory Features Form", "Preconceptional Knowledge and Attitudes Scale", "Preconception Health Behaviours Scale" will be applied.
  The lowest score that can be obtained from the "Preconceptional Knowledge and Attitudes Scale" is 43 and the highest score is 215. As the score obtained from the scale increases, the individual's preconceptional knowledge and attitudes also increase positively.
  The highest score to be obtained from the "Preconception Health Behaviours Scale" is 36 and the lowest score is 0. The high scores obtained from the scale indicate that women's preconceptional period health behaviors are in a positive direction.
Collection of Post-Test Data | Time frame: Four or five months
  The women in the experimental group will be trained according to the health promotion model every week for 8 weeks. The education guide will be prepared by the researcher in line with the literature.The education content will be uploaded to the website and explained by the researcher. After the training is completed, interim test data will be collected in the experimental and control groups. After the training is completed, there will be an 8-week follow-up period and reminders will be given to the women in the experimental group.
  The post-test data of the research is planned to be collected between January 2024 and February 2024. In collecting data, people in the experimental and control groups; "Introductory Features Form", "Preconceptional Knowledge and Attitudes Scale", "Preconception Health Behaviours Scale" will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru BOZCU, Doctorate, Principal Investigator — Erzincan Binali Yildirim Universitesi
Locations (1):
- Erzincan Binali Yıldırım University, Erzincan, Turkey (Türkiye)